CLINICAL TRIAL: NCT00444821
Title: Positive Impact of Endovascular Options for Treating Aneurysms Early (PIVOTAL)
Brief Title: The (PIVOTAL) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis of Primary Endpoint completed
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-2005-01
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: ABDOMINAL AORTIC ANEURYSMS
Keywords: AAA; Aneurysm; AneuRx; Talent
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

ARMS (2):
- Surveillance (No Intervention)
- Early Endovascular Repair (Experimental)
  Interventions: Device: AneuRx AAA stent graft / Talent AAA stent graft

INTERVENTIONS:
Device: AneuRx AAA stent graft / Talent AAA stent graft — Catheter based stent graft inserted to seal off an abdominal aortic aneurysm
  Arms: Early Endovascular Repair

SUMMARY:
The purpose of this study is to compare endovascular repair using any FDA approved Medtronic AAA Stent Graft System versus surveillance in subjects with smaller abdominal aortic aneurysms (AAA)(4-5CM), with respect to AAA rupture and AAA related deaths.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 90 years of age
* Meet all indications for use as stated in the Medtronic Vascular AAA Endograft Instructions for Use
* Maximum aneurysm diameter of 4-5cm
* If female patient with child bearing potential, must have a documented negative pregnancy test within seven(7)days prior to inclusion
* Patient is willing and able to comply with the specified follow-up evaluation
* Life expectancy at least 3 years

Exclusion Criteria:

* Meet any of the Contraindications stated in the Medtronic Vascular AAA Endograft instructions for Use
* Known co-existing condition with a life expectancy of less than 3 years
* Major surgical or interventional procedure (vascular and/or non-vascular)within 30 days prior to study enrollment
* Subjects enrolled in another clinical trial or anticipated to be included into a trial, which may interfere with this study, or subjects already enrolled in this trial before.
* Planned conduit procedure for introduction of endograft

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2005-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ouriel, MD, Principal Investigator — New York Presbyterian Hospital
Locations (65):
- United States (65):
  - University of Alabama, Birmingham, Alabama
  - Tucson Vascular Surgery, Tucson, Arizona
  - University of Arizona - UMC, Tucson, Arizona
  - VA Hospital, Little Rock, Arkansas
  - Palomar Hospital, Escondido, California
  - Long Beach VA Healthcare System, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Stanford University VA, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Leesburg Regional Medical Center, Leesburg, Florida
  - University of South Florida, Tampa, Florida
  - St. Joseph's Research Institute, Atlanta, Georgia
  - Wellstar Clinical Trials, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Adventist Midwest Health, Hinsdale, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Cardiac Surgery Associates, Munster, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Tri-State Vascular Group, Ashland, Kentucky
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Vascular Surgery Associates, Bel Air, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - South Central Regional Medical Center, Laurel, Mississippi
  - St. John's Regional Medical Center, Joplin, Missouri
  - Albany Medical Center, Albany, New York
  - Westchester Medical Center, Hawthorne, New York
  - Columbia University Medical Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Mission / St. Joseph Hospital, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Lindner Clinical Trials Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The Dayton Heart Center, Dayton, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Oregon, Medford, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC Vascular Surgery, Pittsburgh, Pennsylvania
  - North Central Heart Institute, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Heart Hospital, Norfolk, Virginia
  - Sacred Heart Medical Center, Spokane, Washington
  - Wisconsin Heart / Meriter Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Eisenstein EL, Davidson-Ray L, Edwards R, Anstrom KJ, Ouriel K. Economic analysis of endovascular repair versus surveillance for patients with small abdominal aortic aneurysms. J Vasc Surg. 2013 Aug;58(2):302-10. doi: 10.1016/j.jvs.2013.01.038. Epub 2013 Apr 4. PMID 23562339

RESULTS

PARTICIPANT FLOW:
Groups:
- Surveillance: Subjects were assigned to serial ultrasound surveillance
Period: Overall Study
Arm/Group | Surveillance | Early Endovascular Repair
Started | 362 | 366
Received AAA Repair | 122 (Crossed over to AAA repair) | 326 (Underwent AAA repair per protocol)
Completed | 0 | 0
Not Completed | 362 | 366

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surveillance | Early Endovascular Repair | Total
Number analyzed (Participants) | 362 | 366 | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.47 (7.67) | 70.46 (7.80) | 70.46 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 41 | 97
  Male | 306 | 325 | 631
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White race | 343 | 340 | 683
  Hispanic ethnicity | 7 | 7 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 362 | 366 | 728
Baseline AAA size [Mean (Standard Deviation); unit: cm] | 4.45 (0.27) | 4.45 (0.27) | 4.45 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Experienced Rupture or Aneurysm Related Death
Time Frame: 3 years
Population: Study was terminated before all subjects enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance | Early Endovascular Repair
Number analyzed (Participants) | 362 | 366
Participants | 2 | 2

2. Secondary Outcome: Aneurysm Growth >0.5 cm
Description: After repair, AAA enlargement by >0.5cm
Time Frame: 1 year
Population: Study was terminated before all subjects enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance | Early Endovascular Repair
Number analyzed (Participants) | 247 | 263
Participants | 35 | 15

3. Secondary Outcome: Secondary Endovascular Procedures Between the 30-day Post Treatment and 3-year Follow-up
Description: secondary interventions in those that had successful delivery and deployment by treatment group randomized to.
Time Frame: study termination
Population: Study was terminated before all subjects enrolled and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Surveillance | Early Endovascular Repair
Number analyzed (Participants) | 109 | 322
Participants | 5 | 12

ADVERSE EVENTS:
Time Frame: SAEs were collected through study termination and non-SAEs were collected up to and including the 6 month follow-up visit. The mean follow-up was 20 months (range 0-41 months) in each treatment group.
Description: Adverse event is any new, undesirable medial occurrence or change (worsening) of an existing condition in a patient that occurs during treatment, whether or not considered to be associated with the AAA stent graft device.
  Information on all adverse events (serious and non-serious), including deaths, were recorded on the CRFs.
Arm/Group | Surveillance | Early Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 15/362 | 15/366
Serious Adverse Events (participants affected / at risk) | 208/362 | 166/366
Other Adverse Events (participants affected / at risk) | 21/362 | 40/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surveillance (N=362) | Early Endovascular Repair (N=366)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Angina Pectoris (Cardiac disorders) | 2 (2) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 1 (1)
Atrial Fibrillation With Rapid Ventricular Response (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 2 (3)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain Cardiac (Cardiac disorders) | 4 (4) | 1 (2)
Congestive Cardiac Failure Aggravated (Cardiac disorders) | 1 (1) | 1 (2)
Congestive Heart Failure (Cardiac disorders) | 6 (7) | 6 (7)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 6 (6)
Coronary Artery Disease Aggravated (Cardiac disorders) | 3 (3) | 2 (2)
Coronary Artery Disease Progression (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Dilated Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Heart Attack (Cardiac disorders) | 2 (2) | 1 (1)
Heart Block Third Degree (Cardiac disorders) | 0 (0) | 1 (2)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Non St Segment Elevation Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Non-Q Wave Mi (Cardiac disorders) | 6 (6) | 6 (6)
Non-Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Q Wave Mi (Cardiac disorders) | 3 (3) | 2 (2)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Triple Vessel Disease (Cardiac disorders) | 0 (0) | 1 (1)
Unstable Angina (Cardiac disorders) | 4 (4) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Wide Complex Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Benign Positional Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Left) (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Bleeding Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel Ischemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chronic Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohns Disease Aggravated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer Perforated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gerd (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gi Bleed (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 5 (5)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left Lower Quadrant Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mallory Weiss Tear (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea Aggravated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectus Sheath Hematoma (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ruptured Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (2) | 2 (2)
Ugi Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Unspecified Disorder Of Intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Acute Chest Pain (General disorders) | 0 (0) | 1 (1)
Acute Febrile Illness (General disorders) | 0 (0) | 1 (1)
Acute Pain (General disorders) | 0 (0) | 1 (1)
Central Line Complication (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 8 (10) | 7 (10)
Death (General disorders) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Edema Legs (General disorders) | 1 (1) | 0 (0)
Endoleak (General disorders) | 4 (5) | 3 (3)
Fever (General disorders) | 2 (2) | 5 (5)
Fever Of Unknown Origin (General disorders) | 3 (3) | 2 (2)
General Malaise (General disorders) | 2 (2) | 0 (0)
Multiple Organ Failure (General disorders) | 1 (1) | 3 (3)
Nonspecific Chest Pain (General disorders) | 1 (1) | 1 (1)
Stent-Graft Endoleak Type Ii (General disorders) | 0 (0) | 1 (1)
Unspecified Chest Pain (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0)
Acute Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystolithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Common Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic Angioedema (Immune system disorders) | 0 (0) | 1 (1)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (Immune system disorders) | 1 (1) | 0 (0)
Acute Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis Of Arm (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis Of Face (Infections and infestations) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 0 (0) | 1 (1)
Community Acquired Pneumonia (Infections and infestations) | 3 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Groin Abscess (Infections and infestations) | 2 (2) | 1 (1)
Hospital Acquired Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1) | 1 (1)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0)
Mrsa Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 11 (13) | 10 (11)
Post Procedural Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Infection (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (7) | 5 (5)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Surgical Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 4 (4)
Viral Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 3 (3)
Anemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Automobile Accident (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Back Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Broken Leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Closed Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured Sternum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Implantation Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury To Pulmonary Blood Vessel (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration Of Blood Vessel (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar Spine Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 7 (8) | 4 (4)
Wound Oozing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 1 (1) | 3 (3)
Cystoscopy (Investigations) | 0 (0) | 1 (1)
Lung Function Decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hips Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Bulging (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower Extremities Weakness Of (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal Stenosis Cervical (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma Of Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Carcinoma Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Lymphocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal Papillary-Mucinous Carcinoma Of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Melanoma Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Merkel Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Carcinoma Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Cell Carcinoma Of The Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Ganglia Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 4 (4)
Cerebral Bleeding (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Edema (Nervous system disorders) | 1 (1) | 0 (0)
Cva (Nervous system disorders) | 7 (7) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache Recurrent (Nervous system disorders) | 1 (1) | 0 (0)
Intracerebral Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine Headache (Nervous system disorders) | 1 (1) | 0 (0)
Near Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia Lower Limb (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 0 (0)
Pontine Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Tia (Nervous system disorders) | 4 (4) | 2 (2)
Vagal Reaction (Nervous system disorders) | 0 (0) | 1 (1)
Stent-Graft Migration (Product Issues) | 0 (0) | 1 (1)
Anxiety Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety Due To General Medical Condition (Psychiatric disorders) | 5 (5) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-Induced Mood Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 2 (2) | 2 (2)
End Stage Renal Disease (Esrd) (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Artery Occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Disorder Nos (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure Aggravated (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral Calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Voiding Difficulty (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hypertrophy (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Enlarged Prostate (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Copd Exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Respiratory Disorder Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (7)
Subacute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anal Skin Tag Excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic Aneurysm Repair (Surgical and medical procedures) | 5 (5) | 0 (0)
Back Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Catheterization (Surgical and medical procedures) | 1 (1) | 2 (2)
Carotid Endarterectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colostomy Closure (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary Artery Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Craniotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hemodialysis (Surgical and medical procedures) | 0 (0) | 4 (5)
Hernia Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Intubation (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Lung Lobectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Open Reduction Of Fracture (Surgical and medical procedures) | 0 (0) | 1 (1)
Open Reduction Of Fracture With Internal Fixation (Surgical and medical procedures) | 0 (0) | 1 (1)
Pseudophakia (Surgical and medical procedures) | 1 (1) | 0 (0)
Rehabilitation Therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Revision Of Total Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical Intervention (Surgical and medical procedures) | 6 (6) | 4 (4)
Total Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Total Knee Replacement (Surgical and medical procedures) | 4 (4) | 5 (5)
Triple Vessel Bypass Graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular Stent Insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal Aortic Aneurysm (Vascular disorders) | 34 (34) | 1 (1)
Abdominal Aortic Aneurysm Enlargement (Vascular disorders) | 86 (86) | 0 (0)
Acute Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Aneursym (Vascular disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aneurysm Enlargement (Vascular disorders) | 1 (1) | 0 (0)
Aneurysm Ruptured (Vascular disorders) | 1 (1) | 0 (0)
Arterial Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Ascending Aortic Dissection (Vascular disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Vascular disorders) | 4 (4) | 0 (0)
Claudication (Vascular disorders) | 1 (1) | 2 (2)
Dvt (Vascular disorders) | 1 (1) | 2 (2)
Femoral Artery Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Groin Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Iliac Artery Rupture (Vascular disorders) | 1 (1) | 0 (0)
Iliac Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Leg Ischemia (Vascular disorders) | 1 (1) | 0 (0)
Low Blood Pressure (Vascular disorders) | 1 (1) | 0 (0)
Peipheral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 1 (1) | 1 (1)
Popliteal Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Popliteal Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular Disorder (Vascular disorders) | 2 (2) | 5 (5)
Venous Stasis Ulcer (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surveillance (N=362) | Early Endovascular Repair (N=366)
Endoleak (General disorders) | 21 (21) | 40 (47)

LIMITATIONS AND CAVEATS:
Terminated before subjects enrolled & completed follow-up, leading to small numbers. Crossover from the Surveillance Group to Early Endovascular Group led to subjects treated endovascularly being included in the Surveillance Group results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No